CLINICAL TRIAL: NCT02227394
Title: A Double Blind, Double Dummy, Randomized, Two Way Cross-over Study to Compare the Effects of Z7200 and Symbicort® Turbohaler on Functional Respiratory Imaging Parameters in Asthmatic Patients.
Brief Title: Study to Compare the Effects of Z7200 And Symbicort® Turbohaler on Respiratory Imaging Parameters in Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Collaborators: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Z7200K02; 2014-002151-26 (EudraCT Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Asthma; Asthma Chronic; Asthma Bronchial; Asthmatic
Keywords: Asthma; Functional Respiratory Imaging; Computational Fluid Dynamic
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Z7200 - Symbicort® Turbohaler (Experimental): The patients randomized to this sequence were to receive a single dose consisting of 2 inhalations of the test product (Z7200) on the first dosing day (Period 1, Visit 2), then, after a wash out period of at least 3 days but no more of 31 days, a single dose consisting of 2 inhalations of the reference treatment (Symbicort® Turbohaler) on the second dosing day (Period 2, Visit 3).
  Patients were also to receive 2 inhalations with matching placebo to the alternate treatment as a dummy inhaler to achieve double-blinding.
  Z7200 is contained in single dose capsules (HPMC) and it is administered through a single dose dry powder inhaler (DPI), that is structurally correspondent to Aerolizer/Cyclohaler device.
  Strength: Each delivered dose contains budesonide 80 mcg/inhalation and formoterol fumarate dihydrate 2.25 mcg/inhalation; two inhalations (i.e. total dose budesonide/formoterol is 160 mcg/4.5 mcg) to be administered only with the inhaler device (RS-01) provided.
  Interventions: Drug: Z7200; Drug: Symbicort® Turbohaler®
- Symbicort® Turbohaler - Z7200 (Experimental): The patients randomized to this sequence were to receive a single dose consisting of 2 inhalations of the reference treatment (Symbicort® Turbohaler) on the first dosing day (Period 1, Visit 2), then, after a wash out period of at least 3 days but no more of 31 days, a single dose consisting of 2 inhalations of the test product (Z7200) on the second dosing day (Period 2, Visit 3).
  Patients were also to receive 2 inhalations with matching placebo to the alternate treatment as a dummy inhaler to achieve double-blinding.
  Symbicort® Turbohaler® inhalation powder; AstraZeneca UK Limited. Budesonide and formoterol fumarate dihydrate concentration Strength: Each delivered dose contains budesonide 160 mcg/inhalation and formoterol fumarate dihydrate 4.5 mcg/inhalation; two inhalations (i.e. total dose budesonide/formoterol is 320 mcg/9 mcg).
  Interventions: Drug: Z7200; Drug: Symbicort® Turbohaler®

INTERVENTIONS:
Drug: Z7200 — Total dose budesonide/formoterol is 160 mcg/4.5 mcg) to be administered only with the inhaler device (RS-01).
  At visit 2 or 3 (cross-over design)
  Other Names: Test product
Drug: Symbicort® Turbohaler® — Total dose budesonide/formoterol is 320 mcg/9 mcg. At visit 2 or 3 (cross-over design)
  Other Names: Reference product

SUMMARY:
Primary objective:

The primary objective of this study is to evaluate the effect of the products under investigation on functional respiratory imaging parameters and evaluate the particle deposition with Computational fluid dynamics (CFD).

Secondary Objectives:

The secondary objectives of this study were to assess the effect of test product and reference product on:

* lung function (spirometry and body plethysmography),
* exercise capacity (6-Minute Walking Test [6MWT] or equivalent method to measure exercise tolerance),
* dyspnea (Borg Category [C] Ratio [R] 10 [Borg CR10] scale and Visual Analogue Scale [VAS] dyspnea).

Furthermore, the safety of the test product and reference product was evaluated through monitoring of AEs throughout the study.

DETAILED DESCRIPTION:
This study is conducted as a randomized, double blind, double dummy two-period crossover study in stable asthma patients treated in accordance with the Global Initiative for Asthma (GINA) guidelines.

On the first dosing day (Period 1, Visit 2), asthma stability was assessed based on review of pharmacologic treatment monitoring and FEV1 change from the previous visit. Patients were then randomized and allocated to one of two treatment sequences (i.e. test/reference or reference/test). Randomization codes were assigned strictly sequentially as patients became eligible for randomization. Patients received a single dose consisting of two inhalations of either the test product or the reference product, according to the assigned treatment sequence, in the presence of the Investigator or authorized site personnel. In addition, patients received two inhalations with matching placebo to the alternate treatment as a dummy inhaler to achieve double-blinding. All patients followed the same sequence of device inhalation, i.e. Symbicort or placebo Turbohaler first and Z7200 or placebo RS-01 inhaler second.

On the second dosing day (Period 2, Visit 3), patients underwent the same asthma stability check and procedures as in Visit 2. Patients received a single dose consisting of two inhalations of the other treatment (reference in case test product was administered at Visit 2 and vice versa) plus two inhalations with matching placebo to the alternate treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years old.
2. Written informed consent obtained.
3. Patient with a documented diagnosis of asthma according to the Global Initiative for Asthma (GINA) guidelines
4. Patient with a co-operative attitude and ability to correctly use the DPI.
5. Female patient of childbearing potential who confirm that a reliable method of contraception was used at least 14 days before visit 1 and will continue to use a reliable method of contraception during the study, or post-menopausal women (at least 12 months of amenorrhea)
6. Patient must be stable and treated in accordance with the GINA guidelines.
7. Patient must be a non-smoker or ex-smoker who have stopped smoking at least 1 month prior to visit 1 and has a smoking history of < 10 pack years.
8. Patient must be able to understand and complete the protocol requirements, instructions, questionnaires and protocol-stated restrictions.

Exclusion Criteria:

1. Pregnant or lactating female.
2. Unstable patient who developed an asthma exacerbation in the 4 weeks before screening.
3. Patient with upper or lower airways infection in the 4 weeks before screening.
4. Patient unable to perform pulmonary function testing.
5. Patients unable to withdraw fixed combination or long acting bronchodilator inhalation products
6. Patient with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.
7. Patient with active lung cancer or any other chronic disease with poor prognosis and /or affecting patient status.
8. Patient with allergy, sensitivity or intolerance to study drugs and/ or study drug formulation ingredients.
9. Patient unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
10. Patient who received systemic corticosteroids within the last 4 weeks prior to visit
11. Patient who received any investigational new drug within the last 4 weeks prior to visit 1 and is participating in any clinical trial.
12. Patient with a history of alcohol or substance abuse that in the opinion of the investigator may be of clinical significance
13. Patient with diagnosis of Chronic Obstructive Pulmonary Disease (COPD).
14. Patients who has a lactose intolerance or history of allergy to milk proteins.
15. Patients treated with medications or herbal medicines that are strong cytochrome P450 3A4 (CYP3A4) inhibitors (e.g., ritonavir, indinavir, nelfinavir, saquinavir, atazanavir, ketoconazole, itraconazole, voriconazole, fluconazole, cyclosporine, mibefradil, nefazodone, clarithromycin, telithromycin, troleandromycin, norfloxacin, ciprofloxacin) or inducers (e.g. phenobarbital, phenytoin, barbiturates, carbamazepine, oxcarbazepine, rifabutin, rifampin, St John's wort) within 2 weeks prior to Screening Visit and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study procedures were explained to the patients on the screening visit day (Visit 1). Patients who wanted to participate in the study were asked to sign the ICF. Patients were given the chance to ask questions and to clarify their doubts regarding the study either at the screening visit or at any time during the study. Study procedures commenced only after the patient had signed the ICF.
Pre-assignment Details: Only patients who met all inclusion criteria and none of the exclusion criteria were enrolled in the study and entered the run-in period of 7 (minimum) to 31 (maximum) days.
Groups:
- Z7200 - Symbicort® Turbohaler: the patients randomized to this sequence were to receive a single dose consisting of 2 inhalations of the test product (Z7200) on the first dosing day (Period 1, Visit 2), then, after a wash out period of at least 3 days but no more of 31 days, a single dose consisting of 2 inhalations of the reference treatment (Symbicort® Turbohaler) on the second dosing day (Period 2, Visit 3).
  Patients were also to receive 2 inhalations with matching placebo to the alternate treatment as a dummy inhaler to achieve double-blinding.
  Z7200 is contained in single dose capsules (HPMC) and it is administered through a single dose dry powder inhaler (DPI), that is structurally correspondent to Aerolizer/Cyclohaler device.
  Strength: Each delivered dose contains budesonide 80 mcg/inhalation and formoterol fumarate dihydrate 2.25 mcg/inhalation; two inhalations (i.e. total dose budesonide/formoterol is 160 mcg/4.5 mcg) to be administered only with the inhaler device (RS-01) provided.
  Z7200: Total dose budesonide/formoterol is 160 mcg/4.5 mcg) to be administered only with the inhaler device (RS-01).
  At visit 2 or 3 (cross-over design)
  Symbicort® Turbohaler®: Total dose budesonide/formoterol is 320 mcg/9 mcg. At visit 2 or 3 (cross-over design)
- Symbicort® Turbohaler - Z7200: the patients randomized to this sequence were to receive a single dose consisting of 2 inhalations of the reference treatment (Symbicort® Turbohaler) on the first dosing day (Period 1, Visit 2), then, after a washout period of at least 3 days but no more of 31 days, a single dose consisting of 2 inhalations of the test product (Z7200) on the second dosing day (Period 2, Visit 3).
  Patients were also to receive 2 inhalations with a matching placebo to the alternate treatment as a dummy inhaler to achieve double-blinding.
  Symbicort® Turbohaler® inhalation powder; AstraZeneca UK Limited. Budesonide and formoterol fumarate dihydrate concentration Strength: Each delivered dose contains budesonide 160 mcg/inhalation and formoterol fumarate dihydrate 4.5 mcg/inhalation; two inhalations (i.e. total dose budesonide/formoterol is 320 mcg/9 mcg).
  Z7200: Total dose budesonide/formoterol is 160 mcg/4.5 mcg) to be administered only with the inhaler device (RS-01).
  At visit 2 or 3 (cross-over design)
  Symbicort® Turbohaler®: Total dose budesonide/formoterol is 320 mcg/9 mcg. At visit 2 or 3 (cross-over design)
Period: Overall Study
Arm/Group | Z7200 - Symbicort® Turbohaler | Symbicort® Turbohaler - Z7200
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all 20 randomized patients who received at least one dose of study drug.
Groups:
- All Patients: The results of demographic and baseline characteristics are presented for the safety population overall.
Arm/Group | All Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 20

OUTCOME MEASURES:

1. Primary Outcome: Total Airway Volume (iVaw)
Description: The Total Airway Volume is the amount of air that can be inhaled or exhaled during one respiratory cycle. This depicts the functions of the respiratory centers, respiratory muscles and the mechanics of the lung and chest wall. The higher the volume, the better the outcome.
Time Frame: Predose and postdose at the dosing visit V2 [ 7 (minimum) to 31 (maximum) days after Screening] or V3 [ 3 (minimum) to 31(maximum) days after visit 2] up to a maximun of Day 83.
Population: Per-protocol (PP) population: all randomized patients who had correct study drug administration, without any major protocol deviations that could possibly have influenced the assessment of the product effect.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Z7200: Z7200 is contained in single dose capsules (HPMC) and it is administered through a single dose - consisting of two inhalations - dry powder inhaler (DPI), that is structurally correspondent to Aerolizer/Cyclohaler device.
  Strength: Each delivered dose contains budesonide 80 mcg/inhalation and formoterol fumarate dihydrate 2.25 mcg/inhalation; two inhalations (i.e. total dose budesonide/formoterol is 160 mcg/4.5 mcg) to be administered only with the inhaler device (RS-01) provided.
- Symbicort Turbohaler: Symbicort® Turbohaler® inhalation powder; AstraZeneca UK Limited. Budesonide and formoterol fumarate dihydrate concentration Strength: Each delivered dose -- consisting of two inhalations for a total dose budesonide/formoterol is 320 mcg/9 mcg - contains budesonide 160 mcg/inhalation and formoterol fumarate dihydrate 4.5 mcg/inhalation; two inhalations
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
mL
  predose | 49.033 (13.231) | 48.577 (13.430)
  postdose | 51.101 (12.738) | 50.831 (13.478)
  change from predose to postdose | 2.068 (1.659) | 2.255 (2.341)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — The difference between the predose and postdose values of test product and the reference product was compared after applying Benjamini-Hochberg correction (BH) to control the false discovery rate and after Holm-Bonferroni correction (Holm) to control the family-wise error rate; p = 0.727, t-test, 2 sided; Mean Difference (Net) = -0.187, 90% CI 2-sided [-1.098 to 0.724]

2. Primary Outcome: Total Airway Resistance (iRaw)
Description: The Total Airway Resistance refers to degree of resistance to the flow of air through the respiratory tract during inspiration and expiration. The degree of resistance depends on many things, particularly the diameter of the airway and whether flow is laminar or turbulent. The higher the resistance, the worse the outcome.
  In healthy men and women values range between 0.22 to 0.25 kPa/l.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kPas/L
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
kPas/L
  predose | 0.034 (0.016) | 0.037 (0.022)
  postdose | 0.025 (0.011) | 0.026 (0.009)
  change from predose to postdose | -0.008 (0.007) | -0.011 (0.016)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.366, t-test, 2 sided; Mean Difference (Net) = 0.003, 90% CI 2-sided [-0.002 to 0.007]

3. Primary Outcome: Number of Deposited Particles Per Pre-defined Airway Section
Description: To evaluate the particle deposition in the lungs, the Computational Fluid Dynamic (CFD) was used. With CFD, based on the computed tomography (CT) derived geometries of the airways, it is possible to measure the resistance of all airways or subdivisions such as the smaller airways starting from the 3rd bifurcation onwards. The three-dimensional (3D) reconstruction in this CT-based imaging technique allows for an accurate measurement of local volume changes in the central and peripheral airways after the administration of the product. The increased sensitivity of this technique makes it possible to detect changes in airway caliber in early stages of asthma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count of Particles
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 16 | 16
Count of Particles
  Budesonide | 776339324 (111075944) | 17306552 (6985870)
  Formoterol | 80448811 (14821542) | 425671 (179309)

4. Secondary Outcome: Spirometry - FEV1
Description: FEV1 = Forced Expiratory Volume in one second. Forced expiratory volume is the most important measurement of lung function. It measures how much air a person can exhale during a forced breath. The amount of air exhaled may be measured during the first (FEV1), second (FEV2), and/or third seconds (FEV3) of the forced breath.
  Values of between 80% and 120% of the average value are considered normal.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
Liters
  predose | 2.935 (0.904) | 2.905 (0.890)
  postdose | 3.112 (0.896) | 3.058 (0.916)
  change from predose to postdose | 0.178 (0.115) | 0.153 (0.152)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.486, t-test, 2 sided; Mean Difference (Net) = 0.025, 90% CI 2-sided [-0.035 to 0.084]

5. Secondary Outcome: Spirometry - FVC
Description: FVC = Forced Vital Capacity: is the total amount of air exhaled during the FEV test.
  Values of between 80% and 120% of the average value are considered normal.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
Liters
  predose | 4.317 (1.113) | 4.311 (1.125)
  postdose | 4.384 (1.080) | 4.328 (1.155)
  change from predose to postdose | 0.066 (0.173) | 0.018 (0.213)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.413, t-test, 2 sided; Mean Difference (Net) = 0.049, 90% CI 2-sided [-0.052 to 0.150]

6. Secondary Outcome: Spirometry - PEF
Description: PEF = Peak Expiratory Flow: is the maximum flow rate generated during a forceful exhalation, starting from full lung inflation.
  PEF rate primarily reflects large airway flow and depends on the voluntary effort and muscular strength of the patient.
  Normal adult peak expiratory flow ranges between around 400 and 700 liters per minute, although in older it can be lower.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
L/s
  predose | 7.593 (1.978) | 7.465 (1.869)
  postdose | 7.912 (1.948) | 7.883 (1.923)
  change from predose to postdose | 0.319 (0.443) | 0.419 (0.467)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.375, t-test, 2 sided; Mean Difference (Net) = -0.100, 90% CI 2-sided [-0.289 to 0.090]

7. Secondary Outcome: Spirometry - MEF25
Description: MEF25 = Maximal Expiratory Flow at 25% of Forced Vital Capacity (FVC). This parameter is linked to the pathology/obstruction of small airways. Patients with airway obstruction frequently exhibit a marked decrease in MEF25.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
L/s
  predose | 0.700 (0.369) | 0.653 (0.371)
  postdose | 0.873 (0.490) | 0.818 (0.482)
  change from pre-dose to postdose | 0.173 (0.190) | 0.164 (0.221)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.879, t-test, 2 sided; Mean Difference (Net) = 0.009, 90% CI 2-sided [-0.092 to 0.110]

8. Secondary Outcome: Spirometry - MEF50
Description: MEF50 = Maximal Expiratory Flow at 50% of Forced Vital Capacity (FVC). MEF50 is the flow where half of forced vital capacity (FVC) remains to be exhaled. Also this parameter is linked to the pathology/obstruction of small airways. Patients with airway obstruction frequently exhibit a marked decrease in MEF50.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
L/s
  predose | 2.439 (1.151) | 2.350 (1.113)
  postdose | 2.878 (1.265) | 2.767 (1.227)
  change from predose and postdose | 0.440 (0.353) | 0.416 (0.297)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.819, t-test, 2 sided; Mean Difference (Net) = 0.023, 90% CI 2-sided [-0.149 to 0.195]

9. Secondary Outcome: Spirometry - FEV1/FVC Ratio
Description: FEV1/FVC ratio = Tiffeneau Index. It is a calculated ratio use to diagnose obstructive and restrictive lung disease. It represents the proportion of a patient's vital capacity that he/she is able to expire in the first second of forced expiration to the full forced vital capacity. The result of this ratio is expressed as FEV1%.
  Normal values are approximately 75%.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: FEV1%
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
FEV1%
  predose | 67.200 (10.476) | 66.800 (9.600)
  postdose | 70.600 (10.298) | 70.600 (9.484)
  change from predose to postdose | 3.400 (2.927) | 3.800 (2.895)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.643, t-test, 2 sided; Mean Difference (Net) = -0.400, 90% CI 2-sided [-1.870 to 1.070]

10. Secondary Outcome: Body Plethysmography - FRC
Description: FRC = Functional Residual Capacity. It is the volume in the lungs at the end of passive expiration. It is determined by opposing forces of the expanding chest wall and the elastic recoil of the lung. A normal FRC = 1.7 to 3.5 L.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
Liters
  predose | 3.661 (0.765) | 3.685 (0.740)
  postdose | 3.485 (0.707) | 3.498 (0.717)
  change from predose to postdose | -0.176 (0.228) | -0.187 (0.172)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.866, t-test, 2 sided; Mean Difference (Net) = 0.011, 90% CI 2-sided [-0.100 to 0.122]

11. Secondary Outcome: Body Plethysmography - TLC
Description: TLC = Total Lung Capacity. It is the volume of air in the lungs upon the maximum effort of inspiration. Among healthy adults, the average lung capacity is about 6 liters. Age, gender, body composition, and ethnicity are factors affecting the different ranges of lung capacity among individuals.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
Liters
  predose | 7.003 (1.354) | 7.008 (1.458)
  postdose | 7.007 (1.376) | 6.957 (1.447)
  change from predose to postdose | 0.004 (0.151) | -0.051 (0.167)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.346, t-test, 2 sided; Mean Difference (Net) = 0.054, 90% CI 2-sided [-0.043 to 0.152]

12. Secondary Outcome: Body Plethysmography - Raw
Description: Raw = Airway resistance. It is defined as the change in transpulmonary pressure (proximal airway pressure minus the alveolar pressure) required to produce a unit flow of gas through the airways of the lung.
  Are considered as normal all values up to 2.8 kPas/L
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kPas/L
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
kPas/L
  predose | 0.398 (0.419) | 0.411 (0.352)
  postdose | 0.292 (0.266) | 0.276 (0.211)
  change from predose to postdose | -0.106 (0.162) | -0.135 (0.153)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.093, t-test, 2 sided; Mean Difference (Net) = 0.029, 90% CI 2-sided [0.001 to 0.058]

13. Secondary Outcome: Body Plethysmography - SRaw
Description: SRaw = Specific airway resistance: also called volumic airway resistance. sRaw is a corrected index (Raw multiplied by thoracic gas volume) that describes airway behaviour regardless of lung volume. Normal values of sRaw in adult subjects have never been formally defined.
  sRaw is the product of Functional Residual Capacity (FRC) and Airways Resistance (Raw) and can be calculated from the relationship of plethysmographic box pressure (Pbox) to flow during spontaneous breathing.
  sRaw can be derived from the tangent of the slope of box Pressure/Flow. Since Raw has a strong inverse relationship to lung volume, sRaw provides a relatively stable index with which to distinguish effects of disease from those of growth and development. sRaw is significantly increased in asthmatic patients, in those with wheezing disorders, and cystic fibrosis. It has also been shown to be a useful outcome measure for bronchodilator responsiveness studies.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kPas
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
kPas
  predose | 1.656 (1.929) | 1.668 (1.450)
  postdose | 1.137 (1.087) | 1.223 (1.087)
  change from predose to postdose | -0.519 (0.878) | -0.445 (1.066)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.686, t-test, 2 sided; Mean Difference (Net) = -0.074, 90% CI 2-sided [-0.386 to 0.238]

14. Secondary Outcome: Inhalation Profile
Description: The patients' inhalation profile was assessed using a respiration belt. The inhalation profile through device was to be recorded at the moment of study drug administration. Respiratory belts are useful in measuring changes in thoracic or abdominal circumference during respiration. These measurements can indicate inhalation, expiration and breathing strength and can be used to derive breathing rate and characterize breathing patterns
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 16 | 16
Liters | 2.565 (0.829) | 2.366 (1.618)

15. Secondary Outcome: 6MWT
Description: 6MWT = 6 Minutes Walk Test (in meters). The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The longer the walk in that timespan, the better the outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 19 | 19
meters
  predose | 577.789 (69.222) | 583.789 (71.707)
  postdose | 581.789 (72.250) | 598.158 (81.990)
  change from predose to postdose | 4.000 (12.428) | 14.368 (47.174)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.312, t-test, 2 sided; Mean Difference (Net) = -10.368, 90% CI 2-sided [-27.659 to 6.922]

16. Secondary Outcome: Borg CR10 Scale (Pre-6MWT)
Description: Borg category (C) ratio (R) 10 scale = The original Borg CR10 Scale is used to measure the intensity of dyspnoea and fatigue during an exercise (in this case before the walk test). The original one was referred to as a numerical category scale going from 0 to 10. The top of the scale, "0 or nothing at all," means no breathlessness at all.
  The bottom of the scale, "10 or maximal," means the most severe breathlessness that patients have ever experienced or could imagine experiencing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
score on a scale
  predose | 0.805 (1.160) | 0.670 (0.933)
  postdose | 0.935 (1.241) | 0.820 (0.950)
  change from predose to postdose | 0.130 (0.734) | 0.150 (0.511)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.920, t-test, 2 sided; Mean Difference (Net) = -0.020, 90% CI 2-sided [-0.361 to 0.321]

17. Secondary Outcome: Borg CR10 Scale (Post-6MWT)
Description: Borg category (C) ratio (R) 10 scale = The original Borg CR10 Scale is used to measure the intensity of dyspnoea and fatigue during an exercise (in this case after the walk test). The original one was referred to as a numerical category scale going from 0 to 10. The top of the scale, "0 or nothing at all," means no breathlessness at all.
  The bottom of the scale, "10 or maximal," means the most severe breathlessness that patients have ever experienced or could imagine experiencing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
score on a scale
  predose | 1.945 (2.029) | 1.580 (1.265)
  postdose | 1.820 (1.753) | 1.375 (1.290)
  change from pre-dose | -0.125 (1.188) | -0.205 (0.718)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.818, t-test, 2 sided; Mean Difference (Net) = 0.080, 90% CI 2-sided [-0.513 to 0.673]

18. Secondary Outcome: VAS (Pre-6MWT)
Description: VAS = Visual Analogue Scale. A VAS is typically scored by measuring the distance from the bottom of the scale (or left side if oriented horizontally) (In this case before the walk test) to the level indicated by the subject. VAS is typically represented as a vertical or horizontal line, usually 100 millimeters (mm) in length, with descriptors positioned at the extremes of the scale. These extremes go from "not breathless at all"/no shortness of breath" at the bottom or at the far left of the line, to "shortness of breath as bad as can be" on the top or on the right of the line, depending on the patient's opinion.
  measure of the difference in dyspnoea before and after treatment
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
units on a scale | 19.550 (29.416) | 8.150 (25.808)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.034, t-test, 2 sided; Mean Difference (Net) = 11.400, 90% CI 2-sided [2.789 to 20.011]

19. Secondary Outcome: VAS (Post-6MWT)
Description: VAS = Visual Analogue Scale. A VAS is typically scored by measuring the distance from the bottom of the scale (or left side if oriented horizontally) (in this case after the walk test) to the level indicated by the subject. VAS is typically represented as a vertical or horizontal line, usually 100 millimeters (mm) in length, with descriptors positioned at the extremes of the scale. These extremes go from "not breathless at all"/no shortness of breath" at the bottom or at the far left of the line, to "shortness of breath as bad as can be" on the top or on the right of the line, depending on the patient's opinion.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of value
Arm/Group | Z7200 | Symbicort Turbohaler
Number analyzed (Participants) | 20 | 20
percentage of value | 21.450 (23.962) | 15.850 (28.863)
Statistical Analysis 1: Comparison: Z7200 vs Symbicort Turbohaler; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.427, t-test, 2 sided; Mean Difference (Net) = 5.600, 90% CI 2-sided [-6.323 to 17.523]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 2 (Time frame between day 7 and day 31) up to Follow-Up period (at maximum until day 83)
Arm/Group | Z7200 | Symbicort Turbohaler
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Z7200 (N=20) | Symbicort Turbohaler (N=20)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations and Caveats not specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No